CLINICAL TRIAL: NCT05574166
Title: A Phase I Single-Centre, Randomised, Double-Blind, Placebo-Controlled Study in Healthy Volunteers to Evaluate the Safety, Tolerability, and Pharmacokinetics of Escalating Single Doses and Multiple Doses of SP-8356
Brief Title: A Phase I Study to Evaluate Safety and Pharmacokinetics of Escalating Single Doses and Multiple Doses of SP-8356
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Only Part 1 was conducted but not Part 2. Due to the low exposures, definitive safety conclusions could not be made for the targeted exposure levels in the future.
Sponsor: Shin Poong Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SP-8356-1001; 2020-001216-23 (EudraCT Number)
Record Dates: First submitted 2022-10-06; First posted 2022-10-10 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Atherosclerosis; Ischemic Stroke
Keywords: SP-8356; Shinpoong; atherosclerosis; ischaemic stroke
MeSH Terms: conditions — Atherosclerosis; Ischemic Stroke | interventions — SP-8356

STUDY DESIGN:
Intervention Model Description: Dose escalation
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SP-8356 powder (Experimental): Part1 will consist of escalating single doses in five sequential cohorts. Each dose level cohort will consist of 8 subjects: 6 subjects will receive SP-8356 and 2 subjects will receive placebo in fasted state according to the randomization schedule. Subjects in Cohort 3 will receive a single dose of SP-8356 or placebo in the fasted then fed state on separate dosing occasions.
  Interventions: Drug: SP-8356
- Placebo (Placebo Comparator): Part1 will consist of escalating single doses in five sequential cohorts. Each dose level cohort will consist of 8 subjects: 6 subjects will receive SP-8356 and 2 subjects will receive placebo in fasted state according to the randomization schedule. Subjects in Cohort 3 will receive a single dose of SP-8356 or placebo in the fasted then fed state on separate dosing occasions.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SP-8356 — SP-8356 demonstrates anti-atherosclerotic and anti-ischaemic activity as a novel CD147 inhibitor.
  Arms: SP-8356 powder
Drug: Placebo — Placebo for SP-8356 powder
  Arms: Placebo

SUMMARY:
This is a 2-part, single-centre, randomised study in healthy males. Part 1 is a double-blind, randomised, placebo-controlled, single ascending dose (SAD) study in healthy males. Part 2 is a double-blind, randomised, placebo-controlled, multiple ascending dose (MAD) study in healthy males.

DETAILED DESCRIPTION:
2-part, single-centre, randomised study in healthy males. Part 1 is a double-blind, randomised, placebo-controlled, single ascending dose (SAD) study in healthy males. Part 2 is a double-blind, randomised, placebo-controlled, multiple ascending dose (MAD) study in healthy males.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males
2. Aged 18 to 55 years, inclusive, at the time of signing informed consent
3. Body mass index (BMI) of 18.0 to 32.0 kg/m2 as measured at screening
4. Must be willing and able to communicate and participate in the whole study
5. Must provide written informed consent
6. Must agree to adhere to the contraception requirements

Exclusion Criteria:

1. Females
2. Subjects who have received any IMP in a clinical research study within the 90 days prior to the planned first dosing date
3. Subjects who are, or are immediate family members of a study site or sponsor employee
4. Evidence of recent or current SARS-CoV-2 infection. A minimum period of 3 months from resolution of COVID-19 symptoms to dosing must have passed
5. Subjects who have previously been administered IMP in this study.
6. Subjects who have taken part in Part 1 are not permitted to take part in Part 2
7. History of any drug or alcohol abuse in the past 2 years
8. Regular alcohol consumption in males > 21 units per week (1 unit = ½ pint beer, or a 25 mL shot of 40% spirit, 1.5 to 2 Units = 125 mL glass of wine, depending on type)
9. A confirmed positive alcohol breath test at screening or admission
10. Current smokers and those who have smoked within the last 12 months. A confirmed breath carbon monoxide reading of greater than 10 ppm at screening or admission
11. Current users of e-cigarettes and nicotine replacement products and those who have used these products within the last 12 months
12. Subjects who do not have suitable veins for multiple venepunctures/cannulation as assessed by the investigator or delegate at screening
13. Clinically significant abnormal biochemistry, haematology, or urinalysis as judged by the investigator. Subjects with Gilbert's Syndrome are not allowed
14. Subjects that have either a known of family history of QT prolongation or chronic QT prolongation syndrome (i.e. QTc > 450 msec) in repeated ECG
15. Subjects with any clinically significant medical disorders increasing tendency to bleed easily, or having history of recent trauma or surgery, or having history of gout or renal stones
16. Subjects with a clinically significant history of skin disorder such as photosensitivity, eczema or psoriasis.
17. Subjects with a clinically significant history of eye disorders that may affect the interpretation of the ophthalmology assessments as per the judgement of the investigator (only for subjects where ophthalmology assessments will be performed).
18. Confirmed positive drugs of abuse test result
19. Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) or human immunodeficiency virus (HIV) antibody results
20. Evidence of renal impairment at screening, as indicated by an estimated glomerular filtration rate (eGFR) of <80 mL/min/1.73 m2 using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation
21. History of clinically significant cardiovascular, renal, hepatic, chronic respiratory or gastrointestinal disease, neurological or psychiatric disorder, as judged by the investigator
22. Subjects with a history of cholecystectomy or gall stones (Part 1 Cohort 3 only)
23. Serious adverse reaction or serious hypersensitivity to any drug or the formulation excipients
24. Presence or history of clinically significant allergy requiring treatment, as judged by the investigator. Hay fever is allowed unless it is active
25. Donation or loss of greater than 400 mL of blood within the previous 3 months
26. Has a history of photosensitivity or photoallergy
27. Subjects who are taking, or have taken, any prescribed or over-the-counter drug or herbal remedies (other than up to 4 g of paracetamol per day) in the 14 days before IMP administration Exceptions may apply on a case by case basis, if considered not to interfere with the objectives of the study, as determined by the investigator
28. Is taking medication known to cause phototoxic reactions (e.g., tetracyclines, thiazides, nonsteroidal anti-inflammatory drugs) within 4 weeks of enrolling into the study
29. Failure to satisfy the investigator of fitness to participate for any other reason

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2021-01-03 (Actual); Primary Completion 2021-10-28 (Actual); Study Completion 2021-10-29 (Actual)

PRIMARY OUTCOMES:
(Part 1)To investigate the safety and tolerability of single oral doses of SP-8356 in healthy male subjects | up to 3days
  Incidence of adverse events (AEs), and assessment of physical examinations, safety laboratory tests, vital signs, electrocardiograms (ECGs) and ophthalmologic examinations

SECONDARY OUTCOMES:
(Part 1)To characterise the pharmacokinetic (PK) profile of single oral doses of SP-8356 Maximum Observed Drug Concentration (Cmax) | up to 3days
  Evaluate Maximum Observed Drug Concentration (Cmax) of SP-8356.
(Part 1)]To characterise the pharmacokinetic (PK) profile of single oral doses of SP-8356- Area under the plasma concentration versus time curve from time zero to infinity (AUC[0-∞]) | up to 3days
  Evaluate Area Under the Concentration Versus Time Curve from Time Zero to Infinity (AUC[0-∞]) of SP-8356.
(Part 1)To characterise the effect of food on the PK profile of SP-8356 following single oral doses of SP-8356 Maximum Observed Drug Concentration (Cmax) | up to 3days
  Evaluate the effect of food on Maximum Observed Drug Concentration (Cmax) of SP-8356.
(Part 1)To characterise the effect of food on the PK profile of SP-8356 following single oral doses of SP-8356 - Area under the plasma concentration versus time curve from time zero to infinity (AUC[0-∞]) | up to 3days
  Evaluate the effect of food on Area Under the Concentration Versus Time Curve from Time Zero to Infinity (AUC[0-∞]) of SP-8356.

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Mair, MD, PhD, Principal Investigator — Quotient Sciences
Locations (1):
- Quotient Sciences, Nottingham, Mere Way Ruddington Fields Ruddington, United Kingdom

IPD SHARING:
Plan to Share IPD: No